CLINICAL TRIAL: NCT01814072
Title: Opt-IN: Optimization of Remotely Delivered Intensive Lifestyle Treatment for Obesity
Acronym: Opt-IN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Penn State University (Other)
Responsible Party: Principal Investigator, Bonnie Spring, Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIH NIDDK R01DK097364-01; R01DK097364-01 (NIH)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Condition 1 (Experimental): 1) Lifestyle Core; 2) 12 Telephone Coaching Sessions; 3) Report to Primary Care Physician
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician
- Condition 2 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Report to Primary Care Physician; 4) Recommendations to use meal replacements; 5) Buddy training via webinars
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training
- Condition 3 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Report to Primary Care Physician; 4) Regular text messages; 5) Buddy training via webinars
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages; Behavioral: Buddy Training
- Condition 4 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Report to Primary Care Physician; 4) Recommendation to use meal replacements; 5) Regular text messages
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements
- Condition 5 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Buddy training via webinars
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Buddy Training
- Condition 6 (Experimental): 1) Lifestyle Core; 2) 12 telephone coaching sessions; 3) Recommendations to use meal replacements
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Recommendations to use meal replacements
- Condition 7 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Regular text messages
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Text Messages
- Condition 8 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Recommendation to use meal replacements; 4) Regular text messages, 5) Buddy training via webinars
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training
- Condition 9 (Experimental): 1) Lifestyle Core; 2) 24 telephone coaching sessions; 3) Report to Primary Care Physician
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician
- Condition 10 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Report to Primary Care Physician; 4) Recommendation to use meal replacements; 5) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training
- Condition 11 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Report to Primary Care Physician; 4) Regular text messages; 5) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages; Behavioral: Buddy Training
- Condition 12 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Report to Primary Care Physician; 4) Recommendation to use meal replacements; 5) Regular text messages
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements
- Condition 13 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Buddy Training
- Condition 14 (Experimental): 1) Lifestyle Core; 2) 24 telephone coaching sessions; 3) Recommendation to use meal replacements
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Recommendations to use meal replacements
- Condition 15 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Regular text messages
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Text Messages
- Condition 16 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Recommendation to use meal replacements; 4) Regular text messages, 5) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training
- Condition 17 (Experimental): 1) Lifestyle Core; 2) 12 Telephone Coaching Sessions
  Interventions: Behavioral: 12 Telephone Coaching Sessions
- Condition 18 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Recommendations to use meal replacements; 4) Buddy training via webinars
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training
- Condition 19 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Regular text messages; 4) Buddy training via webinars
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Text Messages; Behavioral: Buddy Training
- Condition 20 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Regular text messages; 4) Recommendation to use meal replacements
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements
- Condition 21 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Report to Primary Care Physician; 4) Buddy training via webinars
  Interventions: Behavioral: Report to Primary Care Physician; Behavioral: Buddy Training
- Condition 22 (Experimental): 1) Lifestyle Core; 2) 12 telephone coaching sessions; 3) Report to Primary Care Physician; 4) Recommendations to use meal replacements
  Interventions: Behavioral: Report to Primary Care Physician
- Condition 23 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Report to Primary Care Physician; 4) Regular text messages
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages
- Condition 24 (Experimental): 1) Lifestyle Core; 2) 12 telephone sessions; 3) Report to Primary Care Physician; 4) Recommendation to use meal replacements; 5) Regular text messages, 6) Buddy training via webinars
  Interventions: Behavioral: 12 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training
- Condition 25 (Experimental): 1) Lifestyle Core; 2) 24 telephone coaching sessions
  Interventions: Behavioral: 24 Telephone Coaching Sessions
- Condition 26 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Recommendation to use meal replacements; 4) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training
- Condition 27 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Regular text messages; 4) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Text Messages; Behavioral: Buddy Training
- Condition 28 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Regular text messages; 4) Recommendation to use meal replacements
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements
- Condition 29 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Report to Primary Care Physician; 4) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Buddy Training
- Condition 30 (Experimental): 1) Lifestyle Core; 2) 24 telephone coaching sessions; 3) Report to Primary Care Physician; 4) Recommendation to use meal replacements
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Recommendations to use meal replacements
- Condition 31 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Report to Primary Care Physician; 4) Regular text messages
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages
- Condition 32 (Experimental): 1) Lifestyle Core; 2) 24 telephone sessions; 3) Report to Primary Care Physician; 4) Recommendation to use meal replacements; 5) Regular text messages, 6) Buddy training via webinars
  Interventions: Behavioral: 24 Telephone Coaching Sessions; Behavioral: Report to Primary Care Physician; Behavioral: Text Messages; Behavioral: Recommendations to use meal replacements; Behavioral: Buddy Training

INTERVENTIONS:
Behavioral: 12 Telephone Coaching Sessions — Participants will receive 12 telephone coaching sessions
  Arms: Condition 1; Condition 17; Condition 18; Condition 19; Condition 2; Condition 20; Condition 23; Condition 24; Condition 3; Condition 4; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: 24 Telephone Coaching Sessions — Participants will receive 24 telephone coaching sessions
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 25; Condition 26; Condition 27; Condition 28; Condition 29; Condition 30; Condition 31; Condition 32; Condition 9
Behavioral: Report to Primary Care Physician — Participants will have a report detailing their weight loss progress sent to their primary care physician
  Arms: Condition 1; Condition 10; Condition 11; Condition 12; Condition 2; Condition 21; Condition 22; Condition 23; Condition 24; Condition 29; Condition 3; Condition 30; Condition 31; Condition 32; Condition 4; Condition 9
Behavioral: Text Messages — Participants will receive regular text messages
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 19; Condition 20; Condition 23; Condition 24; Condition 27; Condition 28; Condition 3; Condition 31; Condition 32; Condition 4; Condition 7; Condition 8
Behavioral: Recommendations to use meal replacements — Participants will receive recommendations from their coach to use meal replacements
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 18; Condition 2; Condition 20; Condition 24; Condition 26; Condition 28; Condition 30; Condition 32; Condition 4; Condition 6; Condition 8
Behavioral: Buddy Training — Participants will have a buddy that will be trained via webinars to be a supportive buddy
  Arms: Condition 10; Condition 11; Condition 13; Condition 16; Condition 18; Condition 19; Condition 2; Condition 21; Condition 24; Condition 26; Condition 27; Condition 29; Condition 3; Condition 32; Condition 5; Condition 8

SUMMARY:
The overall objective of the proposed research is to use an innovative methodological framework, the Multiphase Optimization Strategy (MOST), to design, for the first time, an optimized, scalable version of a technology-supported intensive lifestyle intervention (INLI) for obesity. MOST involves highly efficient randomized experimentation to assess the effects of individual treatment components, and thereby identify which components and component levels make important contributions to the overall program effect on weight loss. This information then guides assembly of an optimized treatment package that achieves target outcomes with least resource consumption and participant burden. Because the intervention strategies being tested minimize in-person coaching and leverage technology that participants already own, the new optimized intervention, to be called Opt-IN, will be more scalable than traditional INLIs. Opt-IN will thus enjoy greatly increased reach, and enable significant progress in the fight against obesity.

DETAILED DESCRIPTION:
The goal of the proposed study is to determine the optimal composition of a technology supported intervention for obesity that minimizes expense and burden to participants, while achieving 6 month weight loss outcomes comparable or superior to those achieved by the current full cost, full burden form of INLIs. All intervention components to be examined were selected based on the Opt-IN model's prediction that they enhance behavioral adherence to weight regulation via the designated pathways. The five components to be tested will be: (1) coaching intensity (12 vs. 24 phone sessions), (2) text messaging (No vs. Yes), (3) progress report to participant's primary care provider (No vs. Yes), (4) recommendation to use meal replacements (No vs. Yes), (5) training participants' self-selected buddies to be supportive (No vs. Yes).

ELIGIBILITY:
Inclusion Criteria:

* 18 and 60 years old
* BMI 25-40 kg/m2
* Weight stable (no loss or gain >25 lbs for the past 6 months)
* Not enrolled in any formal weight loss program or taking anti-obesity medications, but interested in losing weight.
* Own a Smartphone and be willing to install the Opt-IN app
* Able to use the app to record dietary intake and weight onto the Smartphone

"Buddy" participants must:

* 18 years of age or older
* Have access to a computer and internet
* Be willing to undergo "Buddy Training" and participate in 4 webinars
* Be willing to provide support and encouragement to the participant

Exclusion Criteria:

* Unstable medical conditions (uncontrolled hypertension, diabetes, unstable angina pectoris, myocardial infarction, transient ischemic attack, cancer undergoing active treatment, or cerebrovascular accident within the past six months)
* History of diabetes requiring insulin supplementation, Crohn's Disease, or a diagnosis of obstructive sleep apnea requiring intervention (i.e. CPAP)
* Use an assistive device for mobility (e.g., wheelchair, walker, cane)
* Plantar fasciitis
* Hospitalization for a psychiatric disorder within the past 5 years
* At risk for adverse cardiovascular (CVD) events with moderate intensity activity
* Cannot read the study questionnaires
* Committed to following an incompatible dietary regimen
* Not be pregnant, trying to get pregnant, or lactating
* Bulimia, binge eating disorder, current substance abuse or dependence (besides nicotine dependence) or report active suicidal ideation
* Low motivation to change
* Cannot live with a current or past Opt-IN participant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 562 (Actual)
Dates: Start 2013-09; Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, Principal Investigator — Northwestern University; Linda Collins, PhD, Principal Investigator — Penn State University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Collins LM, Murphy SA, Strecher V. The multiphase optimization strategy (MOST) and the sequential multiple assignment randomized trial (SMART): new methods for more potent eHealth interventions. Am J Prev Med. 2007 May;32(5 Suppl):S112-8. doi: 10.1016/j.amepre.2007.01.022. PMID 17466815
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Baker TB, Smith SS, Bolt DM, Loh WY, Mermelstein R, Fiore MC, Piper ME, Collins LM. Implementing Clinical Research Using Factorial Designs: A Primer. Behav Ther. 2017 Jul;48(4):567-580. doi: 10.1016/j.beth.2016.12.005. Epub 2017 Jan 7. PMID 28577591
- [Background] Pfammatter AF, Nahum-Shani I, DeZelar M, Scanlan L, McFadden HG, Siddique J, Hedeker D, Spring B. SMART: Study protocol for a sequential multiple assignment randomized controlled trial to optimize weight loss management. Contemp Clin Trials. 2019 Jul;82:36-45. doi: 10.1016/j.cct.2019.05.007. Epub 2019 May 23. PMID 31129369
- [Background] Nahum-Shani I, Dziak JJ, Collins LM. Multilevel factorial designs with experiment-induced clustering. Psychol Methods. 2018 Sep;23(3):458-479. doi: 10.1037/met0000128. Epub 2017 Apr 6. PMID 28383950
- [Background] Terry PE, Brown N, Arnett DK, Cushman M, Spring B, Halpern SD, Burke LE, Grossmeier J, Goetzel R, Lang J, Calitz C, Terry PE, Sanchez E. The Art of Health Promotion ideas for improving health outcomes. Am J Health Promot. 2016 Sep;30(7):563-82. doi: 10.1177/0890117116668866. No abstract available. PMID 27670659
- [Background] Pellegrini CA, Conroy DE, Phillips SM, Pfammatter AF, McFadden HG, Spring B. Daily and Seasonal Influences on Dietary Self-monitoring Using a Smartphone Application. J Nutr Educ Behav. 2018 Jan;50(1):56-61.e1. doi: 10.1016/j.jneb.2016.12.004. PMID 29325663
- [Background] Welch WA, Spring B, Phillips SM, Siddique J. Moderating Effects of Weather-Related Factors on a Physical Activity Intervention. Am J Prev Med. 2018 May;54(5):e83-e89. doi: 10.1016/j.amepre.2018.01.025. Epub 2018 Mar 15. PMID 29551330
- [Background] Burke LE, Ma J, Azar KM, Bennett GG, Peterson ED, Zheng Y, Riley W, Stephens J, Shah SH, Suffoletto B, Turan TN, Spring B, Steinberger J, Quinn CC; American Heart Association Publications Committee of the Council on Epidemiology and Prevention, Behavior Change Committee of the Council on Cardiometabolic Health, Council on Cardiovascular and Stroke Nursing, Council on Functional Genomics and Translational Biology, Council on Quality of Care and Outcomes Research, and Stroke Council. Current Science on Consumer Use of Mobile Health for Cardiovascular Disease Prevention: A Scientific Statement From the American Heart Association. Circulation. 2015 Sep 22;132(12):1157-213. doi: 10.1161/CIR.0000000000000232. Epub 2015 Aug 13. No abstract available. PMID 26271892
- [Background] Piper ME, Cook JW, Schlam TR, Jorenby DE, Smith SS, Collins LM, Mermelstein R, Fraser D, Fiore MC, Baker TB. A Randomized Controlled Trial of an Optimized Smoking Treatment Delivered in Primary Care. Ann Behav Med. 2018 Sep 13;52(10):854-864. doi: 10.1093/abm/kax059. PMID 30212849
- [Background] Booth JN 3rd, Allen NB, Calhoun D, Carson AP, Deng L, Goff DC Jr, Redden DT, Reis JP, Shimbo D, Shikany JM, Sidney S, Spring B, Lewis CE, Muntner P. Racial Differences in Maintaining Optimal Health Behaviors Into Middle Age. Am J Prev Med. 2019 Mar;56(3):368-375. doi: 10.1016/j.amepre.2018.10.020. PMID 30777156
- [Background] Spring B, Pfammatter A, Alshurafa N. First Steps Into the Brave New Transdiscipline of Mobile Health. JAMA Cardiol. 2017 Jan 1;2(1):76-78. doi: 10.1001/jamacardio.2016.4440. No abstract available. PMID 27973672
- [Background] Hoffman SA, Ledford G, Cameron KA, Phillips SM, Pellegrini CA. A qualitative exploration of social and environmental factors affecting diet and activity in knee replacement patients. J Clin Nurs. 2019 Apr;28(7-8):1156-1163. doi: 10.1111/jocn.14719. Epub 2018 Dec 10. PMID 30461097
- [Background] Hekler EB, Michie S, Pavel M, Rivera DE, Collins LM, Jimison HB, Garnett C, Parral S, Spruijt-Metz D. Advancing Models and Theories for Digital Behavior Change Interventions. Am J Prev Med. 2016 Nov;51(5):825-832. doi: 10.1016/j.amepre.2016.06.013. PMID 27745682
- [Background] Kheirkhahan M, Tudor-Locke C, Axtell R, Buman MP, Fielding RA, Glynn NW, Guralnik JM, King AC, White DK, Miller ME, Siddique J, Brubaker P, Rejeski WJ, Ranshous S, Pahor M, Ranka S, Manini TM. Actigraphy features for predicting mobility disability in older adults. Physiol Meas. 2016 Oct;37(10):1813-1833. doi: 10.1088/0967-3334/37/10/1813. Epub 2016 Sep 21. PMID 27653966
- [Background] Collins LM, Kugler KC, Gwadz MV. Optimization of Multicomponent Behavioral and Biobehavioral Interventions for the Prevention and Treatment of HIV/AIDS. AIDS Behav. 2016 Jan;20 Suppl 1(0 1):S197-214. doi: 10.1007/s10461-015-1145-4. PMID 26238037
- [Background] Piper ME, Schlam TR, Cook JW, Smith SS, Bolt DM, Loh WY, Mermelstein R, Collins LM, Fiore MC, Baker TB. Toward precision smoking cessation treatment I: Moderator results from a factorial experiment. Drug Alcohol Depend. 2017 Feb 1;171:59-65. doi: 10.1016/j.drugalcdep.2016.11.025. Epub 2016 Nov 25. PMID 28013098
- [Background] Piper ME, Fiore MC, Smith SS, Fraser D, Bolt DM, Collins LM, Mermelstein R, Schlam TR, Cook JW, Jorenby DE, Loh WY, Baker TB. Identifying effective intervention components for smoking cessation: a factorial screening experiment. Addiction. 2016 Jan;111(1):129-41. doi: 10.1111/add.13162. Epub 2015 Nov 19. PMID 26582269
- [Background] Collins LM, Dziak JJ, Kugler KC, Trail JB. Factorial experiments: efficient tools for evaluation of intervention components. Am J Prev Med. 2014 Oct;47(4):498-504. doi: 10.1016/j.amepre.2014.06.021. Epub 2014 Aug 1. PMID 25092122
- [Background] Spring B, Pellegrini CA, Pfammatter A, Duncan JM, Pictor A, McFadden HG, Siddique J, Hedeker D. Effects of an abbreviated obesity intervention supported by mobile technology: The ENGAGED randomized clinical trial. Obesity (Silver Spring). 2017 Jul;25(7):1191-1198. doi: 10.1002/oby.21842. Epub 2017 May 11. PMID 28494136
- [Background] Pellegrini CA, Pfammatter AF, Conroy DE, Spring B. Smartphone applications to support weight loss: current perspectives. Adv Health Care Technol. 2015 Jul;1:13-22. doi: 10.2147/AHCT.S57844. PMID 26236766
- [Background] Spring B, Ockene JK, Gidding SS, Mozaffarian D, Moore S, Rosal MC, Brown MD, Vafiadis DK, Cohen DL, Burke LE, Lloyd-Jones D; American Heart Association Behavior Change Committee of the Council on Epidemiology and Prevention, Council on Lifestyle and Cardiometabolic Health, Council for High Blood Pressure Research, and Council on Cardiovascular and Stroke Nursing. Better population health through behavior change in adults: a call to action. Circulation. 2013 Nov 5;128(19):2169-76. doi: 10.1161/01.cir.0000435173.25936.e1. Epub 2013 Oct 7. No abstract available. PMID 24100544
- [Background] Baker TB, Collins LM, Mermelstein R, Piper ME, Schlam TR, Cook JW, Bolt DM, Smith SS, Jorenby DE, Fraser D, Loh WY, Theobald WE, Fiore MC. Enhancing the effectiveness of smoking treatment research: conceptual bases and progress. Addiction. 2016 Jan;111(1):107-16. doi: 10.1111/add.13154. Epub 2015 Nov 19. PMID 26581974
- [Background] Pellegrini CA, Hoffman SA, Daly ER, Murillo M, Iakovlev G, Spring B. Acceptability of smartphone technology to interrupt sedentary time in adults with diabetes. Transl Behav Med. 2015 Sep;5(3):307-14. doi: 10.1007/s13142-015-0314-3. PMID 26327936
- [Background] Piper ME, Cook JW, Schlam TR, Smith SS, Bolt DM, Collins LM, Mermelstein R, Fiore MC, Baker TB. Toward precision smoking cessation treatment II: Proximal effects of smoking cessation intervention components on putative mechanisms of action. Drug Alcohol Depend. 2017 Feb 1;171:50-58. doi: 10.1016/j.drugalcdep.2016.11.027. Epub 2016 Nov 24. PMID 28013097
- [Background] Schlam TR, Fiore MC, Smith SS, Fraser D, Bolt DM, Collins LM, Mermelstein R, Piper ME, Cook JW, Jorenby DE, Loh WY, Baker TB. Comparative effectiveness of intervention components for producing long-term abstinence from smoking: a factorial screening experiment. Addiction. 2016 Jan;111(1):142-55. doi: 10.1111/add.13153. Epub 2015 Nov 19. PMID 26581819
- [Background] Watkins E, Newbold A, Tester-Jones M, Javaid M, Cadman J, Collins LM, Graham J, Mostazir M. Implementing multifactorial psychotherapy research in online virtual environments (IMPROVE-2): study protocol for a phase III trial of the MOST randomized component selection method for internet cognitive-behavioural therapy for depression. BMC Psychiatry. 2016 Oct 6;16(1):345. doi: 10.1186/s12888-016-1054-8. PMID 27716200
- [Background] Collins LM, Nahum-Shani I, Almirall D. Optimization of behavioral dynamic treatment regimens based on the sequential, multiple assignment, randomized trial (SMART). Clin Trials. 2014 Aug;11(4):426-434. doi: 10.1177/1740774514536795. Epub 2014 Jun 5. PMID 24902922
- [Background] Cook JW, Collins LM, Fiore MC, Smith SS, Fraser D, Bolt DM, Baker TB, Piper ME, Schlam TR, Jorenby D, Loh WY, Mermelstein R. Comparative effectiveness of motivation phase intervention components for use with smokers unwilling to quit: a factorial screening experiment. Addiction. 2016 Jan;111(1):117-28. doi: 10.1111/add.13161. Epub 2015 Nov 19. PMID 26582140
- [Background] Pellegrini CA, Hoffman SA, Collins LM, Spring B. Optimization of remotely delivered intensive lifestyle treatment for obesity using the Multiphase Optimization Strategy: Opt-IN study protocol. Contemp Clin Trials. 2014 Jul;38(2):251-9. doi: 10.1016/j.cct.2014.05.007. Epub 2014 May 17. PMID 24846621
- [Background] Pellegrini CA, Hoffman SA, Collins LM, Spring B. Corrigendum to "Optimization of remotely delivered intensive lifestyle treatment for obesity using the Multiphase Optimization Strategy: Opt-IN study protocol" [Contemp. Clin. Trials 38 (2014) 251-259]. Contemp Clin Trials. 2015 Nov;45(Pt B):468-469. doi: 10.1016/j.cct.2015.09.001. Epub 2015 Nov 29. No abstract available. PMID 28802730
- [Derived] Spring B, Pfammatter AF, Marchese SH, Stump T, Pellegrini C, McFadden HG, Hedeker D, Siddique J, Jordan N, Collins LM. A Factorial Experiment to Optimize Remotely Delivered Behavioral Treatment for Obesity: Results of the Opt-IN Study. Obesity (Silver Spring). 2020 Sep;28(9):1652-1662. doi: 10.1002/oby.22915. Epub 2020 Jul 12. PMID 32656994
- [Derived] Pfammatter AF, Marchese SH, Pellegrini C, Daly E, Davidson M, Spring B. Using the Preparation Phase of the Multiphase Optimization Strategy to Develop a Messaging Component for Weight Loss: Formative and Pilot Research. JMIR Form Res. 2020 May 13;4(5):e16297. doi: 10.2196/16297. PMID 32347804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8593 were screened. 1159 attended orientation. 1078 signed consent. 562 were randomized.
Pre-assignment Details: Participants who signed an informed consent were invited to attend a baseline assessment where they were screened further for entry and exclusion criteria. Baseline data was gathered. Participants who continued to be eligible were scheduled for the randomization session where they learned their study assignment.
Groups:
- 1. 12 Calls, PCP: Participant's received biweekly (12) coaching calls, and PCP Reports
- 2. 12 Calls, PCP, MR, Buddy: Participant's received biweekly (12) coaching calls, PCP Reports, Meal Replacement Recommendations, and Buddy Training.
- 3. 12 Calls, PCP, Texts, Buddy: Participant received 12 calls, PCP Reports, Texts, and Buddy Training
- 4. 12 Calls, PCP, Texts, MR: Participant received 12 calls, PCP Reports, Texts, and Meal Replacement Recommendations
- 5. 12 Calls, Buddy: Participant received 12 calls, and Buddy Training
- 6. 12 Calls, MR: Participant received 12 calls, and Meal Replacement Recommendations
- 7. 12 Calls, Texts: Participant received 12 calls, and Texts
- 8. 12 Calls, Texts, MR, Buddy: Participant received 12 calls, Texts, Meal Replacement Recommendations, and Buddy Training
- 9. 24 Calls, PCP: Participants received 24 calls, and PCP Reports
- 10. 24 Calls, PCP, MR, Buddy: Participants received 24 calls, PCP Reports, Meal Replacement Recommendations, and Buddy Training
- 11. 24 Calls, PCP, Texts, Buddy: Participants received 24 calls, PCP Reports, Texts, and Buddy Training
- 12. 24 Calls, PCP, Texts, MR: Participants received 24 calls, PCP Reports, Texts, and Meal Replacement Recommendations
- 13. 24 Calls, Buddy: Participants received 24 calls, and Buddy Training
- 14. 24 Calls, MR: Participants received 24 calls, and Meal Replacement Recommendations
- 15. 24 Calls, Texts: Participants received 24 calls, and Texts
- 16. 24 Calls, Texts, MR, Buddy: Participants received 24 calls, Texts, Meal Replacement Recommendations, and Buddy Training
- 17. 12 Calls: Participants received 12 calls
- 18. 12 Calls, MR, Buddy: Participants received 12 calls, Meal Replacement Recommendations, and Buddy Training
- 19. 12 Calls, Texts, Buddy: Participants received 12 calls, Texts, and Buddy Training
- 20. 12 Calls, Texts, MR: Participants received 12 calls, Texts, Meal Replacement Recommendations
- 21. 12 Calls, PCP, Buddy: Participants received 12 calls, PCP Reports, and Buddy Training
- 22. 12 Calls, PCP, MR: Participants received 12 calls, PCP Reports, and Meal Replacement Recommendations
- 23. 12 Calls PCP, Texts: Participants received 12 calls, PCP Reports, and Texts
- 24. 12 Calls, PCP, Texts, MR, Buddy: Participants received 12 calls, PCP Reports, Texts, Meal Replacement Recommendations, and Buddy Training
- 25. 24 Calls: Participants received 24 calls
- 26. 24 Calls, MR, Buddy: Participants received 24 calls, Meal Replacement Recommendations, and Buddy Training
- 27. 24 Calls, Texts, Buddy: Participants received 24 calls, Texts, and Buddy Training
- 28. 24 Calls, Texts, MR: Participants received 24 calls, Texts, and Meal Replacement Recommendations
- 29. 24 Calls, PCP, Buddy: Participants received 24 calls, PCP Reports, and Buddy Training
- 30. 24 Calls, PCP, MR: Participants received 24 calls, PCP Reports, and Meal Replacement Recommendations
- 31. 24 Calls, PCP, Texts: Participants received 24 calls, PCP Reports, and Texts
- 32. 24 Calls, PCP, Texts, MR, Buddy: Participants received 24 calls, PCP Reports, Texts, Meal Replacement Recommendations, and Buddy Training
Period: Overall Study
Arm/Group | 1. 12 Calls, PCP | 2. 12 Calls, PCP, MR, Buddy | 3. 12 Calls, PCP, Texts, Buddy | 4. 12 Calls, PCP, Texts, MR | 5. 12 Calls, Buddy | 6. 12 Calls, MR | 7. 12 Calls, Texts | 8. 12 Calls, Texts, MR, Buddy | 9. 24 Calls, PCP | 10. 24 Calls, PCP, MR, Buddy | 11. 24 Calls, PCP, Texts, Buddy | 12. 24 Calls, PCP, Texts, MR | 13. 24 Calls, Buddy | 14. 24 Calls, MR | 15. 24 Calls, Texts | 16. 24 Calls, Texts, MR, Buddy | 17. 12 Calls | 18. 12 Calls, MR, Buddy | 19. 12 Calls, Texts, Buddy | 20. 12 Calls, Texts, MR | 21. 12 Calls, PCP, Buddy | 22. 12 Calls, PCP, MR | 23. 12 Calls PCP, Texts | 24. 12 Calls, PCP, Texts, MR, Buddy | 25. 24 Calls | 26. 24 Calls, MR, Buddy | 27. 24 Calls, Texts, Buddy | 28. 24 Calls, Texts, MR | 29. 24 Calls, PCP, Buddy | 30. 24 Calls, PCP, MR | 31. 24 Calls, PCP, Texts | 32. 24 Calls, PCP, Texts, MR, Buddy
Started | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 19 | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 17 | 18 | 17 | 16 | 16 | 17 | 17 | 18 | 17 | 16 | 18 | 17 | 18 | 17 | 17 | 17
3-mo Visit | 15 | 18 | 16 | 18 | 15 | 15 | 16 | 18 | 18 | 15 | 18 | 17 | 16 | 16 | 16 | 16 | 16 | 16 | 14 | 13 | 15 | 17 | 15 | 18 | 13 | 14 | 17 | 14 | 15 | 16 | 16 | 17
Intent to Treat | 4 | 2 | 3 | 0 | 4 | 6 | 4 | 1 | 3 | 5 | 1 | 2 | 3 | 2 | 3 | 2 | 3 | 1 | 3 | 5 | 2 | 1 | 4 | 1 | 6 | 2 | 2 | 4 | 4 | 3 | 2 | 0
Completed | 14 | 16 | 15 | 18 | 14 | 12 | 14 | 17 | 16 | 13 | 17 | 16 | 15 | 16 | 15 | 16 | 14 | 17 | 14 | 11 | 14 | 16 | 13 | 17 | 11 | 14 | 16 | 13 | 14 | 14 | 15 | 17
Not Completed | 4 | 2 | 3 | 0 | 4 | 6 | 4 | 1 | 3 | 5 | 1 | 2 | 3 | 2 | 3 | 2 | 3 | 1 | 3 | 5 | 2 | 1 | 4 | 1 | 6 | 2 | 2 | 4 | 4 | 3 | 2 | 0
Not completed — Lost to Follow-up | 2 | 2 | 2 | 0 | 2 | 3 | 3 | 1 | 2 | 3 | 1 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 3 | 3 | 2 | 1 | 3 | 1 | 4 | 1 | 1 | 2 | 3 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants (562).
Groups:
- 1. 12 Calls, PCP: Participants received biweekly (12) coaching calls, and PCP Reports
- 2. 12 Calls, PCP, MR, Buddy: Participants received biweekly (12) coaching calls, PCP Reports, Meal Replacement Recommendations, and Buddy Training.
- 3. 12 Calls, PCP, Texts, Buddy: Participants received 12 calls, PCP Reports, Texts, and Buddy Training
- 4. 12 Calls, PCP, Texts, MR: Participants received 12 calls, PCP Reports, Texts, and Meal Replacement Recommendations
- 5. 12 Calls, Buddy: Participants received 12 calls, and Buddy Training
- 6. 12 Calls, MR: Participants received 12 calls, and Meal Replacement Recommendations
- 7. 12 Calls, Texts: Participants received 12 calls, and Texts
- 8. 12 Calls, Texts, MR, Buddy: Participants received 12 calls, Texts, Meal Replacement Recommendations, and Buddy Training
- Total: Total of all reporting groups
Arm/Group | 1. 12 Calls, PCP | 2. 12 Calls, PCP, MR, Buddy | 3. 12 Calls, PCP, Texts, Buddy | 4. 12 Calls, PCP, Texts, MR | 5. 12 Calls, Buddy | 6. 12 Calls, MR | 7. 12 Calls, Texts | 8. 12 Calls, Texts, MR, Buddy | 9. 24 Calls, PCP | 10. 24 Calls, PCP, MR, Buddy | 11. 24 Calls, PCP, Texts, Buddy | 12. 24 Calls, PCP, Texts, MR | 13. 24 Calls, Buddy | 14. 24 Calls, MR | 15. 24 Calls, Texts | 16. 24 Calls, Texts, MR, Buddy | 17. 12 Calls | 18. 12 Calls, MR, Buddy | 19. 12 Calls, Texts, Buddy | 20. 12 Calls, Texts, MR | 21. 12 Calls, PCP, Buddy | 22. 12 Calls, PCP, MR | 23. 12 Calls PCP, Texts | 24. 12 Calls, PCP, Texts, MR, Buddy | 25. 24 Calls | 26. 24 Calls, MR, Buddy | 27. 24 Calls, Texts, Buddy | 28. 24 Calls, Texts, MR | 29. 24 Calls, PCP, Buddy | 30. 24 Calls, PCP, MR | 31. 24 Calls, PCP, Texts | 32. 24 Calls, PCP, Texts, MR, Buddy | Total
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 19 | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 17 | 18 | 17 | 16 | 16 | 17 | 17 | 18 | 17 | 16 | 18 | 17 | 18 | 17 | 17 | 17 | 562
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (8.6) | 43.2 (14.2) | 41.7 (10.9) | 40.2 (11.2) | 31.4 (9.1) | 40.5 (9.9) | 40.8 (12.2) | 39.4 (12.9) | 39.5 (8.3) | 38.7 (8.9) | 39.1 (11.2) | 40.6 (12.0) | 40.4 (9.1) | 36.3 (10.6) | 39.8 (12.8) | 35.8 (11.8) | 38.2 (12.0) | 39.2 (10.5) | 37.4 (10.9) | 32.2 (7.1) | 36.7 (6.0) | 40.3 (10.8) | 40.1 (11.6) | 37.9 (12.8) | 35.7 (9.6) | 47.3 (10.2) | 35.1 (9.0) | 41.0 (10.1) | 39.1 (11.7) | 37.2 (9.9) | 40.6 (12.8) | 39.9 (12.0) | 38.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 16 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 14 | 14 | 14 | 12 | 13 | 14 | 14 | 14 | 14 | 13 | 14 | 14 | 14 | 14 | 13 | 13 | 459
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 4 | 3 | 4 | 4 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 16 | 11 | 15 | 18 | 16 | 13 | 16 | 16 | 18 | 17 | 13 | 17 | 17 | 17 | 13 | 16 | 12 | 14 | 13 | 14 | 15 | 16 | 15 | 16 | 18 | 14 | 16 | 15 | 15 | 17 | 489
  Not Hispanic or Latino | 4 | 0 | 1 | 4 | 3 | 0 | 1 | 2 | 3 | 2 | 0 | 1 | 4 | 1 | 0 | 0 | 4 | 2 | 3 | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 0 | 2 | 2 | 2 | 1 | 0 | 53
  Unknown or Not Reported | 2 | 0 | 1 | 3 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 10 | 15 | 11 | 12 | 16 | 15 | 15 | 10 | 15 | 14 | 14 | 12 | 12 | 15 | 15 | 14 | 13 | 15 | 9 | 14 | 11 | 14 | 12 | 14 | 12 | 13 | 14 | 9 | 13 | 10 | 13 | 16 | 417
  Black | 3 | 3 | 4 | 3 | 2 | 2 | 1 | 5 | 4 | 3 | 4 | 4 | 5 | 2 | 3 | 3 | 1 | 2 | 3 | 1 | 2 | 1 | 4 | 3 | 1 | 1 | 3 | 5 | 4 | 2 | 2 | 1 | 87
  Asian | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 16
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other/Unknown | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 3 | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 5 | 1 | 0 | 36
Weight (kg) [Mean (Standard Deviation); unit: Kilograms] | 88.9 (10.6) | 91.2 (14.0) | 87.3 (12.0) | 88.8 (14.0) | 90.4 (11.3) | 90.0 (13.3) | 97.8 (13.3) | 87.3 (13.4) | 94.4 (14.7) | 93.1 (12.9) | 97.6 (14.4) | 88.1 (13.4) | 89.6 (12.9) | 87.2 (13.9) | 94.3 (14.7) | 91.3 (11.3) | 88.4 (13.7) | 90.2 (15.2) | 90.8 (14.8) | 83.3 (9.8) | 92.9 (14.8) | 86.1 (10.5) | 98.0 (15.3) | 90.5 (17.6) | 80.7 (12.2) | 89.8 (9.9) | 90.1 (12.0) | 85.5 (10.8) | 89.7 (13.4) | 93.7 (16.6) | 86.8 (11.5) | 86.1 (16.0) | 90.0 (13.6)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change (kg) From Baseline to Month 6, Main Effect of Time
Description: Estimated mean change from Baseline to Month 6 were obtained from a linear mixed models analysis of variance to account for missing data. All randomized participants were utilized in the model (ITT analysis).
Time Frame: From Baseline to Month 6
Population: ITT population: all randomized participants with at least one weight value. The decision to analyze all randomized participants together for aim 1, rather than separately by arm, was pre-specified in the the Protocol/Statistical Analysis Plan for the purposes of assessing the main effect of time.
Measure: Mean (95% Confidence Interval); unit: Kg
Groups:
- All Reporting Groups: All participants regardless of individual randomly assigned combination of On- or Off switched levels of all intervention factors, weight measured at baseline and at Month 6.
Arm/Group | All Reporting Groups
Number analyzed (Participants) | 562
Kg | -4.8 [-5.3 to -4.4]
Statistical Analysis 1: Comparison: All Reporting Groups; Test type: Superiority; p < .001, Mixed Models Analysis

2. Primary Outcome: Weight Change (kg) From Baseline to Month 6, Time by Factor Interaction
Description: Estimated mean change from Baseline to Month 6 were obtained from a linear mixed models analysis of variance to account for missing data. All randomized participants were utilized in the model (ITT analysis).
  This outcome measure is reported as an additional effect beyond that of Outcome Measure 1 (each component has it's own weight loss effect that is above and beyond the weight change calculated in the Outcome Measure 1 analyses).
Time Frame: From Baseline to Month 6
Population: ITT population: all randomized participants with at least one weight value.
Measure: Mean (95% Confidence Interval); unit: Kg
Groups:
- Coaching Calls: 12 bi-weekly coaching calls (Off) or 24 weekly coaching calls (On)
- PCP Reports: Participant's primary care physician was (On) or was not (Off) sent a progress report after the 3 and 6 month assessments.
- Text Messages: Participants either received (On) or did not receive (Off) push notifications through the app at their preferred time or when they opened the app.
- Meal Replacements: Participants either received (On) or did not receive (Off) a one week supply of meal replacement bars and shakes. Those who did receive a 1-week supply of meal replacements were provided with recommendations on each coaching call to continue using these products throughout the intervention.
- Buddy Training: Participant buddies either received (On) or did not receive (Off) additional training.
Arm/Group | Coaching Calls | PCP Reports | Text Messages | Meal Replacements | Buddy Training
Number analyzed (Participants) | 562 | 562 | 562 | 562 | 562
Kg | .1244 [-.3026 to .5513] | -.0226 [-.4495 to .4044] | .0840 [-.3429 to .5109] | .1081 [-.3188 to .5350] | -.4353 [-.8622 to -.0084]
Statistical Analysis 1: Comparison: Coaching Calls; Test type: Superiority; p = 0.567, Mixed Models Analysis; Estimated Change = 0.1244, 95% CI 2-sided [-.3026 to .5513]
Statistical Analysis 2: Comparison: PCP Reports; Test type: Superiority; p = 0.917, Mixed Models Analysis; Estimated Change = -0.0226, 95% CI 2-sided [-.4495 to .4044]
Statistical Analysis 3: Comparison: Text Messages; Test type: Superiority; p = 0.699, Mixed Models Analysis; Estimated Change = 0.084, 95% CI 2-sided [-.3429 to .5109]
Statistical Analysis 4: Comparison: Meal Replacements; Test type: Superiority; p = 0.619, Mixed Models Analysis; Estimated Change = 0.1081, 95% CI 2-sided [-.3188 to .5350]
Statistical Analysis 5: Comparison: Buddy Training; Test type: Superiority; p = 0.046, Mixed Models Analysis; Estimated Change = -0.4353, 95% CI 2-sided [-.8622 to -.0084]

3. Secondary Outcome: Intervention for <$500
Description: Using the results from primary aim 1, an intervention with only active treatment components with the largest treatment effect that can be obtained for implementation costs of $500 or less was identified and built.
Time Frame: 6 months
Population: ITT population: weight loss data from all randomized participants with at least one weight value; combined with cost data for study implementation (staff time, supplies, etc.)
Measure: Number; unit: dollars
Groups:
- All Reporting Groups: All participants regardless of individual randomly assigned combination of On- or Off switched levels of all intervention factors.
Arm/Group | All Reporting Groups
Number analyzed (Participants) | 562
dollars | 427
Statistical Analysis 1: Comparison: All Reporting Groups; Using the results from primary aim 1, an intervention with only active treatment components with the largest treatment effect that can be obtained for implementation costs of $500 or less was identified and built; Test type: Other; p = 0.051, Mixed Models Analysis; Estimated Change = 0.424, 95% CI 2-sided [-0.002 to 0.850]

4. Other Pre Specified Outcome: Treatment Adherence
Description: Treatment adherence is a hypothesized mediator that will be operationalized as the number of treatment sessions completed divided by the number of treatment sessions offered (12 or 24)
Time Frame: 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Self-monitoring Adherence
Description: Self-monitoring is a hypothesized mediator that will be operationalized as the number of days recording weight, dietary intake, and physical activity
Time Frame: 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Self-efficacy
Description: Self-efficacy is an exploratory mediator that will be assessed to examine treatment effects on confidence about performing two categories of behaviors associated with weight loss: diet and physical activity
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Self-Regulation
Description: Self-regulation is an exploratory mediator that will be assessed using the Three Factor Eating Questionnaire and Treatment Self-Regulation Questionnaire
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Supportive Accountability
Description: Supportive accountability is an exploratory mediator that will be measured by assessing two constructs that define supportive accountability: therapeutic alliance and perceived autonomy support
Time Frame: 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Facilitation
Description: Facilitation is an exploratory mediator that will be measured by rating how much the tools provided by the study have changed their environment and by the Weight Management Support Inventory
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from randomization to 6-month follow-up. All 562 participants in the study were enrolled between 2013 and 2017.
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16 | Condition 17 | Condition 18 | Condition 19 | Condition 20 | Condition 21 | Condition 22 | Condition 23 | Condition 24 | Condition 25 | Condition 26 | Condition 27 | Condition 28 | Condition 29 | Condition 30 | Condition 31 | Condition 32
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/19 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/17 | 0/18 | 0/17 | 0/16 | 0/16 | 0/17 | 0/17 | 0/18 | 0/17 | 0/16 | 0/18 | 0/17 | 0/18 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 1/18 | 0/18 | 0/18 | 0/18 | 0/19 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 1/18 | 0/17 | 0/18 | 0/17 | 0/16 | 0/16 | 0/17 | 0/17 | 0/18 | 0/17 | 0/16 | 0/18 | 0/17 | 0/18 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 6/18 | 8/18 | 7/18 | 4/18 | 4/18 | 2/18 | 5/18 | 8/18 | 8/18 | 8/18 | 4/18 | 9/18 | 7/18 | 8/18 | 8/18 | 8/18 | 5/17 | 2/18 | 1/17 | 2/16 | 2/16 | 2/17 | 1/17 | 2/18 | 3/17 | 2/16 | 3/18 | 4/17 | 3/18 | 2/17 | 3/17 | 1/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition 1 (N=18) | Condition 2 (N=18) | Condition 3 (N=18) | Condition 4 (N=18) | Condition 5 (N=18) | Condition 6 (N=18) | Condition 7 (N=18) | Condition 8 (N=18) | Condition 9 (N=19) | Condition 10 (N=18) | Condition 11 (N=18) | Condition 12 (N=18) | Condition 13 (N=18) | Condition 14 (N=18) | Condition 15 (N=18) | Condition 16 (N=18) | Condition 17 (N=17) | Condition 18 (N=18) | Condition 19 (N=17) | Condition 20 (N=16) | Condition 21 (N=16) | Condition 22 (N=17) | Condition 23 (N=17) | Condition 24 (N=18) | Condition 25 (N=17) | Condition 26 (N=16) | Condition 27 (N=18) | Condition 28 (N=17) | Condition 29 (N=18) | Condition 30 (N=17) | Condition 31 (N=17) | Condition 32 (N=17)
Brain bleed (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant slipped and fell on tile floor, hit his head and suffered severe concussion and brain bleeding. Was cleared for full activity after a month of recovery.
severe head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — sustained a severe head injury in a car accident, unable to complete study activities
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition 1 (N=18) | Condition 2 (N=18) | Condition 3 (N=18) | Condition 4 (N=18) | Condition 5 (N=18) | Condition 6 (N=18) | Condition 7 (N=18) | Condition 8 (N=18) | Condition 9 (N=18) | Condition 10 (N=18) | Condition 11 (N=18) | Condition 12 (N=18) | Condition 13 (N=18) | Condition 14 (N=18) | Condition 15 (N=18) | Condition 16 (N=18) | Condition 17 (N=17) | Condition 18 (N=18) | Condition 19 (N=17) | Condition 20 (N=16) | Condition 21 (N=16) | Condition 22 (N=17) | Condition 23 (N=17) | Condition 24 (N=18) | Condition 25 (N=17) | Condition 26 (N=16) | Condition 27 (N=18) | Condition 28 (N=17) | Condition 29 (N=18) | Condition 30 (N=17) | Condition 31 (N=17) | Condition 32 (N=17)
thyroid imbalance (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
thyroid cancer (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
anterior scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
stomach ache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
stomach ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
medication switch (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bicycle accident (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — bicycle accident, no injury
neutropenia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
food poisoning (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
sinus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
strep throat (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
common cold (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
stomach flu (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
staph infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
general respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
intolerance to meal replacements (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bladder cancer (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
skin cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pinched nerve (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
seizure disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
spinal stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
polycystic ovary syndrome (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abnormal mammogram (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — doctor monitoring, no official diagnosis
uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
breast cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
degenerative disc disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
capsulitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dental procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
skin surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
foot surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hyperhidrosis surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
stomach surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
elbow surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
kidney stone surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
lasik eye surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
muscle soreness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
blisters (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
joint soreness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ankle sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
migraine (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
muscle cramps (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
knee sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
mild concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT01814072/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT01814072/ICF_001.pdf